CLINICAL TRIAL: NCT04921540
Title: Etude Comparative Multicentrique Prospective évaluant la Prise en Charge Chirurgicale associée à Une cautérisation Chimique Par Acide TCA Par Rapport à la Prise en Charge Chirurgicale Standard Dans le Traitement de l'Ongle incarné
Brief Title: Ingrown Toenails : Surgery Only Versus Surgery + Chemical Cauterization With TCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-090
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2020-07

CONDITIONS: Relapse; Quality of Life; Complication; Pain, Postoperative
Keywords: Ingrown nail; Simple surgery; Surgery with chemical cauterisation; Trichloroacetic acid; Relapse; Quality of life
MeSH Terms: conditions — Recurrence; Pain, Postoperative; Nails, Ingrown | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermatologic intervention (Experimental): Surgery with chemical cauterisation TCA
  Interventions: Procedure: Ingrown toenails with surgery with chemical cauterisation
- Orthopedic intervention (Active Comparator): Only surgery
  Interventions: Procedure: Ingrown toenails with only surgery

INTERVENTIONS:
Procedure: Ingrown toenails with surgery with chemical cauterisation — Removal of the ingrown lateral part of the toenail and chemical cauterisation
  Arms: Dermatologic intervention
Procedure: Ingrown toenails with only surgery — Removal of the ingrown lateral part of the toenail with directed Healing pad
  Arms: Orthopedic intervention

SUMMARY:
Ingrown toenail is a very common disease in the general population that touches young adults. There are lots of treatments from local care of pedicure to surgery with matricectomy. Gold standard of symptomatic and painful ingrown toenail is the simple surgery with matricectomy and with suture or directed healing pad.

For many years chemical cauterisation with phenolic acid is used, a method with very few relapses and with a more simple pad. However, because of a lack of information about this phenolic acid, the pharmaceutical laboratory withdrew it from the market.

The new method to replace phenolic acid is trichloroacetic acid, used mainly in cosmetics for peeling. This method was already compared to phenolic acid and showed equal results with fewer laps of application and a low cost. The comparison between acid trichloroacetic method and the gold standard surgery was never done and will be the goal of this study.

It's an open, non randomised, comparative, multicentric (2 centers) study with two groups : common surgery and surgery with chemical cauterisation For this study the investigators will compare between the two groups : gain of quality of life at one month after surgery, difference of pain between before, one week and one month after surgery, the occurrence of adverse events and number of relapses at one year.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ingrown toenail
* Patient informed and with signed informed consent

Exclusion Criteria:

* Medical history of ingrown toenail on the concerned nail
* Other nail disease
* Pregnancy
* Allergy to local anesthetic or to trichloroacetic acid

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Relapses | one year
  Relapses of ingrown toenail on the operated nail

SECONDARY OUTCOMES:
Gain of quality of life | Baseline and one month after the surgery
  Quality of life will be measured with the Dermatology Life Quality Index adapted to the nail, there are 9 questions that will be filled by the patient. Each questions have 4 possibilities to 0 (no problem) to 3(hugely). So the score go to 0 to 27.
  Questions are, on last 7 days :
  * Did your nail itch, burn or hurt you ?
  * Did you feel embarrassed or complexed by your nail ?
  * Did you have problem to go shopping, to do the housework ?
  * Did you have problem to put on your shoes?
  * Did your nail problem affect your hobbies and activity ?
  * Did you have problem to do sport ?
  * Did your nail embarrased you in your job or your studies ?
  * Did your nail complicate your relationship's with your friends, parents or spouse?
  * Did your nail deteriorate your sexual life ?
Complications | At one week and one month after surgery
  Bleeding, infection, pain
Pain on the nail | Baseline, one week and one month after surgery
  Pain report on a numeric scale of pain to 0 (no pain) to 10(worst pain possible)
Time before restart sport | Restart sport at one month yes/no
  Time to recover a normal physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Pr DOMPMARTIN ANNE, Study Director — CHU CAEN
Locations (2):
- France (2):
  - Centre hospitalier universitaire de CAEN, Caen, Normandy
  - Centre hospitalier Mémorial France Etats Unis, Saint-Lô, Normandy

IPD SHARING:
Plan to Share IPD: No